CLINICAL TRIAL: NCT02826291
Title: Sentinel Lymph Node Mapping in Endometrial Cancer Patients Combined With One-step Nucleic Acid Amplification (OSNA)
Brief Title: SLNM in Endometrial Cancer Combined With OSNA
Acronym: SLNM/OSNA
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: University Hospital Pilsen (Other)
Responsible Party: Principal Investigator, Jan Kosťun, MUDr., Charles University, Czech Republic
Other Study IDs: OSNA-EC-01
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Endometrial Cancer
Keywords: OSNA; sentinel; lymph; node; endometrial; cancer
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of the tissue homogenate will be retained and may be used for further testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RD-100i, OSNA: SLNM and OSNA assessment of sentinel lymph nodes compared to ultrastaging
  Interventions: Device: RD-100i, OSNA

INTERVENTIONS:
Device: RD-100i, OSNA — quantitative reverse transcription polymerase chain reaction (qRT-PCR) cytokeratin-19 detection in specimen (sentinel lymph node)

SUMMARY:
The aim of the study is to compare one-step nucleic acid amplification method (OSNA) with histological ultrastaging examination in the sentinel lymph node assessment in patients with endometrial cancer.

The molecular biologic method OSNA is a modern way of metastatic spread detection in lymphatic nodes using quantitative reverse transcription polymerase chain reaction. Cytokeratin 19 (CK 19) was selected based on previous studies as the optimal mRNA marker (detected by OSNA).

The intraoperative identification and rapid assessment of sentinel lymph nodes by OSNA could help to improve the standards of care in endometrial cancer patients.

DETAILED DESCRIPTION:
Method:

After the sentinel lymph node detection (ICG, 99m Tc or Bleu Patente) and sentinel node/nodes removal is performed, the node/nodes is/are cut in 2-mm slices parallel to short axis of the node. The odd-numbered blocks will be examined by the OSNA method and the even-numbered blocks will be examined by conventional histopathological methods including immunohistochemistry.

Statistical analysis to identify differences will be performed subsequently.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial cancer
* Signed informed consent

Exclusion Criteria:

* Inclusion criteria not met
* Pregnant patients
* Patients participating in other clinical studies
* Patients who have been judged to be an inappropriate candidate by any medical care provider

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years diagnosed with endometrial cancer.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-03; Primary Completion 2018-01-31 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
number of CK 19 copies detected by OSNA | 14 days
  Number of CK 19 copies will be assessed: 250-5000 micrometastasis, more than 5000 copies macrometastasis. This result will be compared to histological ultrastaging examination.

CONTACTS AND LOCATIONS:
Overall Officials: Ondřej Topolčan, Prof. MUDr., Study Chair — Department of Nuclear Medicine, Medical School and Teaching Hospital in Pilsen, Charles University in Prague, Prague, Czech Republic; Zdeněk Novotný, Doc.MUDr., Study Chair — Department of Obstetrics and Gynaecology, University Hospital in Pilsen, Charles University in Prague, Czech Republic
Locations (1):
- Faculty Hospital in Pilsen, Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagai T, Niikura H, Okamoto S, Nakabayashi K, Matoda M, Utsunomiya H, Nagase S, Watanabe M, Takeshima N, Yaegashi N. A new diagnostic method for rapid detection of lymph node metastases using a one-step nucleic acid amplification (OSNA) assay in endometrial cancer. Ann Surg Oncol. 2015 Mar;22(3):980-6. doi: 10.1245/s10434-014-4038-2. Epub 2014 Sep 5. PMID 25190122
- [Background] Yamamoto H, Sekimoto M, Oya M, Yamamoto N, Konishi F, Sasaki J, Yamada S, Taniyama K, Tominaga H, Tsujimoto M, Akamatsu H, Yanagisawa A, Sakakura C, Kato Y, Matsuura N. OSNA-based novel molecular testing for lymph node metastases in colorectal cancer patients: results from a multicenter clinical performance study in Japan. Ann Surg Oncol. 2011 Jul;18(7):1891-8. doi: 10.1245/s10434-010-1539-5. Epub 2011 Feb 3. PMID 21290195
- [Background] Okamoto S, Niikura H, Nakabayashi K, Hiyama K, Matoda M, Takeshima N, Watanabe M, Nagase S, Otsuki T, Yaegashi N. Detection of sentinel lymph node metastases in cervical cancer: assessment of KRT19 mRNA in the one-step nucleic acid amplification (OSNA) method. Gynecol Oncol. 2013 Sep;130(3):530-6. doi: 10.1016/j.ygyno.2013.06.027. Epub 2013 Jun 28. PMID 23811115
- [Background] Buglioni S, Di Filippo F, Terrenato I, Casini B, Gallo E, Marandino F, Maini CL, Pasqualoni R, Botti C, Di Filippo S, Pescarmona E, Mottolese M. Quantitative molecular analysis of sentinel lymph node may be predictive of axillary node status in breast cancer classified by molecular subtypes. PLoS One. 2013;8(3):e58823. doi: 10.1371/journal.pone.0058823. Epub 2013 Mar 22. PMID 23533593
- [Background] Mariani A, Webb MJ, Keeney GL, Podratz KC. Routes of lymphatic spread: a study of 112 consecutive patients with endometrial cancer. Gynecol Oncol. 2001 Apr;81(1):100-4. doi: 10.1006/gyno.2000.6111. PMID 11277658
- [Background] Colombo N, Creutzberg C, Amant F, Bosse T, Gonzalez-Martin A, Ledermann J, Marth C, Nout R, Querleu D, Mirza MR, Sessa C; ESMO-ESGO-ESTRO Endometrial Consensus Conference Working Group. ESMO-ESGO-ESTRO Consensus Conference on Endometrial Cancer: Diagnosis, Treatment and Follow-up. Int J Gynecol Cancer. 2016 Jan;26(1):2-30. doi: 10.1097/IGC.0000000000000609. PMID 26645990
- [Background] Kim CH, Soslow RA, Park KJ, Barber EL, Khoury-Collado F, Barlin JN, Sonoda Y, Hensley ML, Barakat RR, Abu-Rustum NR. Pathologic ultrastaging improves micrometastasis detection in sentinel lymph nodes during endometrial cancer staging. Int J Gynecol Cancer. 2013 Jun;23(5):964-70. doi: 10.1097/IGC.0b013e3182954da8. PMID 23694985
- [Background] Leitao MM Jr, Khoury-Collado F, Gardner G, Sonoda Y, Brown CL, Alektiar KM, Hensley ML, Soslow RA, Barakat RR, Abu-Rustum NR. Impact of incorporating an algorithm that utilizes sentinel lymph node mapping during minimally invasive procedures on the detection of stage IIIC endometrial cancer. Gynecol Oncol. 2013 Apr;129(1):38-41. doi: 10.1016/j.ygyno.2013.01.002. Epub 2013 Jan 12. PMID 23321065